CLINICAL TRIAL: NCT05674188
Title: The Physiologic and Emotional Effects of Augmented Reality Simulation Versus In Person Simulation - A Noninferiority, Randomized Controlled Trial
Brief Title: AR vs In Person Simulation for Medical Workplace Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 68663
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Augmented Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality Enhanced Simulation (Treatment group) (Experimental): Participants will experience augmented simulations with a holographic mixed-reality setting based on different workplace scenarios such as medical error and workplace harassment via Augmented Reality (AR) headset.
  Interventions: Behavioral: Augmented Reality Headset
- Traditional In Situ Simulation (Control group) (No Intervention): Participants will experience in-person simulations of different workplace scenarios such as medical error and workplace harassment

INTERVENTIONS:
Behavioral: Augmented Reality Headset — Augmented simulation of workplace-related scenarios of pre-recorded videos using the same actors
  Arms: Augmented Reality Enhanced Simulation (Treatment group)

SUMMARY:
This study will evaluate the physiologic and emotional effects of an augmented reality (AR) simulation versus an in-person simulation. This is a single institution, non-inferiority, randomized controlled trial. The target enrollment will be 100 participants in each group for a total of 200 participants. One group will wear an AR headset and participate in an AR medical crisis scenario and the other group will participate in the same scenario with a traditional, mannequin based in situ simulation.

ELIGIBILITY:
Inclusion Criteria:

* Hospital providers, including nurses, physician assistants, physicians, physician trainees, and other healthcare workers at Lucile Packard Children's Hospital (LPCH) and affiliated facilities who communicate with patients daily will be included

Exclusion Criteria:

* Participants with reported severe motion sickness
* Nausea
* Seizure disorder
* Currently using chronotropic heart medications, such as β blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Parasympathetic response indexed by RSA | Duration of simulation (15-20 minutes)
  Measured via respiratory sinus arrhythmia (RSA) in hertz using chest biometric sensors in 30-second epochs.

SECONDARY OUTCOMES:
Sytem Usability Scale (SUS) | Post-simulation (5 minutes)
  10-item questionnaire with a scale from 1- 5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale to measure usability. Only administered to the AR group.
ISO 9241-400 | Post-simulation (5 minutes)
  6-item ergonomic questionnaire with a scale from 1- 5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale only administered to the AR group.
Simulation Design Scale (SDS) | Post-simulation (5-10 minutes)
  20-item questionnaire with a scale from 1- 5, 1 being strongly disagree to 5 being strongly agree on a five-point Likert scale to assess user satisfaction
Learning effectiveness | 5 months-post simulation (5 minutes)
  Five months post-simulation, an assessment was sent out to participants with a 10-item, multiple choice with questions related to key learning points about resuscitation management.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Caruso, MD, MEd, Principal Investigator — clinical professor
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rama A, Rojas-Pino MS, Wang EY, Rodriguez ST, Suen MY, Titzler JS, Zuniga-Hernandez M, Jackson C, Rosales O, Collins F, Caruso TJ. The Physiologic Effect of Augmented Reality Simulation Versus Traditional Simulation: A Noninferiority, Randomized Controlled Trial. J Educ Perioper Med. 2025 Apr 8;27(1):E740. doi: 10.46374/VolXXVII_Issue1_Rama. eCollection 2025 Jan-Mar. PMID 40207076